CLINICAL TRIAL: NCT00727311
Title: Treatment of Chronic Hepatitis C With PegIntron Injector and Rebetol (Post Marketing Surveillance Study)
Brief Title: Real-life Surveillance Study of Patients With Chronic Hepatitis C Treated With PegIntron Injector and Rebetol (Study P04538)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04538
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PegIntron + Rebetol: Participants with chronic hepatitis C, who are either treatment-naïve or previously relapsed after receiving interferon monotherapy
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031) injector; Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) injector — PegIntron administered at a dose 1.5 μg/kg/week, according to the Summary of Product Characteristics (SPC) and approved European labeling
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered at a dose of 800-1200 mg/day (on a weight-basis) according to the SPC and approved European labeling
  Other Names: SCH 18908

SUMMARY:
The objective of the study is to assess the safety and efficacy of PegIntron injector and Rebetol administered to participants with chronic hepatitis C. Participants will be treated by general practitioners in clinical practice as part of the post-marketing surveillance study. The study will assess the rates of eradication of the hepatits C virus and the rates of serious adverse events reported with PegIntron (1.5 μg/kg/week) and Rebetol (800-1200 mg/day) in common medical practice in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic hepatitis C
* At least 18 years old
* Treatment-naïve or relapse to interferon monotherapy
* Platelets >= 100,000/mm^3
* Neutrophil counts >= 1,500/ mm^3
* Thyroid Stimulating Hormone (TSH) must be within normal limits
* Hemoglobin >= 12 gr/dl (females); >= 13 gr/dl (males)
* Intravenous drug abusers (Ex-IVDA) participants being under stable substitution for at least 6 months
* Women of childbearing potential must have a routine pregnancy test performed monthly during treatment and for 7 months thereafter. Sexually active female participants of childbearing potential must be practicing adequate contraception (intrauterine device, oral contraceptives, implanted contraceptives, surgical sterilization, barrier method, or monogamous relationship with a male partner who has had a vasectomy or is using a condom (+ spermicide) during the treatment period and for 7 months after stopping treatment
* Sexually active male participants must be practicing acceptable methods of contraception (vasectomy, use of condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 7 months after stopping treatment

Exclusion Criteria:

* Contraindications as per the SPC and approved European labeling
* Hypersensitivity to the active substance or to any inteferons or to any of the excipients
* Pregnant woman
* Woman who are breast-feeding
* Existence of or history of severe psychiatric condition, in particular severe depression, suicidal ideation or suicide attempt
* A history of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous six months
* Severe debilitating medical conditions, including participants with chronic renal failure or creatinine clearance < 50 mL/min
* Autoimmune hepatitis or history of autoimmune disease
* Severe hepatic dysfunction or decompensated cirrhosis of the liver
* Pre-existing thyroid disease unless it can be controlled with conventional therapy
* Epilepsy and/or compromised central nervous system function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic hepatitis C, who are either treatment-naïve or previous relapsers after interferon monotherapy, from 500 sites in Germany
Sampling Method: Non-Probability Sample
Enrollment: 2302 (Actual)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- PegIntron + Rebetol: Participants with chronic hepatitis C, who are either treatment-naïve or previously relapsed after receiving interferon monotherapy. PegIntron was administered at a dose 1.5 μg/kg/week, according to the Summary of Product Characteristics (SPC) and approved European labeling.
  Rebetol was administered at a dose of 800-1200 mg/day (on a weight-basis) according to the SPC and approved European labeling.
Period: Overall Study
Arm/Group | PegIntron + Rebetol
Started | 2302
Completed | 1195
Not Completed | 1107
Not completed — Did not receive drug | 316
Not completed — Missing end of therapy data | 205
Not completed — Adverse Event | 58
Not completed — Lack of Efficacy | 242
Not completed — Lost to Follow-up | 73
Not completed — Withdrawal by Subject | 77
Not completed — Other | 97
Not completed — Multiple reasons | 39

BASELINE CHARACTERISTICS:
Arm/Group | PegIntron + Rebetol
Number analyzed (Participants) | 2302
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age was for the evaluable population of 1986 participants.
  years | 42.1 (11.7)
Sex/Gender, Customized [Number; unit: participants]
  Male | 1169
  Female | 766
  Gender information not captured | 367
Region of Enrollment [Number; unit: participants]
  Germany | 2302

OUTCOME MEASURES:

1. Primary Outcome: Number of Hepatitis C Virus Ribonucleic Acid (HCV-RNA) Negative Participants at End of Therapy (EoT)
Description: HCV-RNA level was measured by polymerase chain reaction (PCR).
Time Frame: 24 weeks in genotypes 2 and 3, and 48 weeks in genotypes 1, 4, 5, and 6
Population: Number of evaluable participants at EoT
Measure: Number; unit: Participants
Arm/Group | PegIntron + Rebetol
Number analyzed (Participants) | 1781
Participants | 1306

2. Primary Outcome: Number of Participants With Early Virologic Response (EVR)
Description: EVR was defined as at least a 2 log reduction in HCV-RNA or HCV-RNA
  negativity from baseline to Week 12
Time Frame: Treatment Week 12
Population: Number of evaluable participants at 12 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | PegIntron + Rebetol
Number analyzed (Participants) | 1823
Participants | 1168

3. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR)
Description: SVR was defined as HCV-RNA negativity at EoT and at the follow-up 6 months after the EoT
Time Frame: 24 weeks post-treatment (Week 48 or 72, depending on genotype)
Population: Number of evaluable participants with follow-up information
Measure: Number; unit: Participants
Arm/Group | PegIntron + Rebetol
Number analyzed (Participants) | 1986
Participants | 888

4. Primary Outcome: Number of HCV-RNA Negative Participants at Follow-up
Description: HCV-RNA was measured by PCR.
Time Frame: 24 weeks post-treatment (Weeks 48 or 72, depending on genotype)
Population: Number of participants with results at the 6 month follow-up examination
Measure: Number; unit: Participants
Arm/Group | PegIntron + Rebetol
Number analyzed (Participants) | 1616
Participants | 887

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 58/2302
Other Adverse Events (participants affected / at risk) | 151/2302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2302)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5)
LEUKOPENIA (Blood and lymphatic system disorders) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (3)
PALPITATIONS (Cardiac disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 2 (2)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 5 (5)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1)
ADVERSE EVENT (General disorders) | 1 (1)
ASTHENIA (General disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
ENANTHEMA (General disorders) | 1 (1)
FATIGUE (General disorders) | 5 (5)
INJECTION SITE INFLAMMATION (General disorders) | 2 (2)
INJECTION SITE PRURITUS (General disorders) | 1 (1)
MALAISE (General disorders) | 1 (1)
PYREXIA (General disorders) | 2 (2)
HYPERSENSITIVITY (Immune system disorders) | 2 (2)
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
SEPSIS (Infections and infestations) | 1 (1)
UROSEPSIS (Infections and infestations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
BLOOD COUNT (Investigations) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2)
RED BLOOD CELL COUNT DECREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 4 (4)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
CEREBELLAR INFARCTION (Nervous system disorders) | 1 (1)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3)
HYPOTONIA (Nervous system disorders) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1)
AGGRESSION (Psychiatric disorders) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1)
DEPENDENCE (Psychiatric disorders) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 4 (4)
DEPRESSION (Psychiatric disorders) | 1 (1)
LISTLESS (Psychiatric disorders) | 1 (1)
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 1 (1)
MIDDLE INSOMNIA (Psychiatric disorders) | 1 (1)
MOOD SWINGS (Psychiatric disorders) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2302)
FATIGUE (General disorders) | 151 (158)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All rights according to the results belong to Essex, Germany. Publications or transmission of data need a previous written agreement of the company.